CLINICAL TRIAL: NCT00712335
Title: The Effects of Montelukast on Sputum Cells and Inflammatory Markers in Smokers With Asthma
Brief Title: The Effects of Montelukast on Smokers With Asthma
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Inje University (Other)
Responsible Party: Principal Investigator, Chang-Keun Kim, Dr., Director, Asthma and Allergy Center; Chairman of Pediatrics; Professor of Pediatrics, Inje University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: MASK2008
Record Dates: First submitted 2008-07-07; First posted 2008-07-09 (Estimated); Results first posted 2012-05-16 (Estimated); Last update posted 2012-05-16 (Estimated); Status verified 2012-04

CONDITIONS: Asthmatic Smokers; Non-asthmatic Smokers
Keywords: asthmatics; smokers; inhaled corticosteroids; leukotriene receptor antagonists
MeSH Terms: conditions — Asthma | interventions — Fluticasone; montelukast; Leukotriene Antagonists; Salmeterol Xinafoate

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- 1 (Experimental): Asthmatic smokers treated with combination therapy:
  Fluticasone propionate dosage - DPI 250 mcg BID for 3 months Salmeterol dosage - DPI 50 mcg BID for 3 months
  Interventions: Drug: Fluticasone Propionate; Drug: Salmeterol
- 2 (Experimental): Asthmatic smoker treated with Montelukast only:
  Montelukast dosage: PO 10 mg QHS for 3 months
  Interventions: Drug: Montelukast
- 3 (Active Comparator): Non-smoking asthmatics treated with combination therapy:
  Fluticasone propionate dosage - DPI 250 mcg BID for 3 months Salmeterol dosage - DPI 50 mcg BID for 3 months
  Interventions: Drug: Fluticasone Propionate; Drug: Salmeterol
- 4 (Active Comparator): Non-smoking asthmatic treated with Montelukast only:
  Montelukast dosage: PO 10 mg QHS for 3 months
  Interventions: Drug: Montelukast
- 5 (No Intervention): Normal controls

INTERVENTIONS:
Drug: Fluticasone Propionate — DPI 250 mcg BID for 3 weeks
  Other Names: inhaled corticosteroid
  Arms: 1; 3
Drug: Montelukast — PO 10 mg QHS for 3 weeks
  Other Names: leukotriene receptor antagonist
  Arms: 2; 4
Drug: Salmeterol — DPI 50mg BID for 3 weeks
  Other Names: long-acting beta-agonist
  Arms: 1; 3

SUMMARY:
The purpose of this study is:

1. To compare neutrophilia, eosinophilic inflammatory markers and asthma symptom indices between smokers and non-smokers.
2. To elucidate the mechanism by which cigarette smokers are resistant to corticosteroids.

DETAILED DESCRIPTION:
Many smokers have insufficient control of their symptoms due to inefficacy of ICS in this subpopulation of asthmatics. Cigarette smoking has been shown to stimulate production of cysLTs. CysLTs could activate production of IL-8 for neutrophilia as well as cause eosinophilia in the airway of asthmatics.

LTRAs are felt to be less efficacious than ICS in smokers with asthma. However, LTRA's unique mechanism of action could be particularly efficacious in preventing worsening symptoms and lung function for smokers with asthma. Given this, along with the fact that ICS are less effective in smokers, targeting cysLT could lead to significant clinical benefits for asthmatic smokers.

Data from this study may possibly serve as crucial data for the significant clinical benefits for asthmatic smokers and determination of the mechanism of corticosteroid resistance in smokers with asthma.

ELIGIBILITY:
Inclusion Criteria:

Asthmatics:

* clinical history of asthma for at least 1 year
* with evidence of reversible airway obstruction,
* two documented FEV1 between 60-85%,
* PC20 < 4mg/ml by methacholine challenge test
* and average baseline β-agonist use of 2 puffs/day

Smokers:

* smoke 1/2 to 2 packs a day
* with a smoking history of 5-30 pack years

Non-smokers:

* Non-smokers will have either never smoked or have stopped smoking cigarettes over 5 years ago

Exclusion Criteria:

* positive HCG (for females)
* have a respiratory tract infection or need oral corticosteroids within the preceding 6 weeks
* history of COPD or respiratory disorder other than asthma
* history of psychiatric illness
* allergy to fluticasone propionate, salmeterol, montelukast or any of their components
* significant, unstable medical condition other than asthma
* history of life-threatening asthma exacerbation requiring intubation and mechanical ventilation in the last ten years

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 105 (Actual)
Dates: Start 2007-02; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chang-Keun Kim, MD, PhD, Principal Investigator — Asthma and Allergy Center, Inje University Sanggye Paik Hospital
Locations (1):
- Asthma and Allergy Center, Inje University Sanggye Paik Hospital, Seoul, South Korea

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period: January 2008-April 2011 Recruitment location: Asthma and Allergy Center, Inje University Sanggye Paik Hospital
Pre-assignment Details: After randomization, a 10-day washout period followed in which subjects were taken off all medications except albuterol metered dose inhaler as needed. After the washout period, baseline induced sputum was obtained in each group along with primary and secondary endpoints. This was followed by a 3-week run in period.
Groups:
- Asthmatic Smokers Treated With Combination Therapy: Asthmatic smokers treated with combination therapy:
  Fluticasone propionate dosage - DPI 250 mcg BID for 3 months Salmeterol dosage - DPI 50 mcg BID for 3 months
- Asthmatic Smoker Treated With Montelukast Only: Asthmatic smoker treated with Montelukast only:
  Montelukast dosage - PO 10 mg QHS for 3 months
- Non-smoking Asthmatic Treated With Combination Therapy: Non-smoking asthmatic treated with combination therapy:
  Fluticasone propionate dosage - DPI 250 mcg BID for 3 months Salmeterol dosage - DPI 50 mcg BID for 3 months
- Non-smoking Asthmatic Treated With Montelukast Only: Non-smoking asthmatic treated with Montelukast only:
  Montelukast dosage - PO 10 mg QHS for 3 months
- Normal Controls: Normal controls did not receive any treatment.
Period: Overall Study
Arm/Group | Asthmatic Smokers Treated With Combination Therapy | Asthmatic Smoker Treated With Montelukast Only | Non-smoking Asthmatic Treated With Combination Therapy | Non-smoking Asthmatic Treated With Montelukast Only | Normal Controls
Started | 8 | 32 | 11 | 24 | 30
Completed | 5 | 15 | 6 | 19 | 30
Not Completed | 3 | 17 | 5 | 5 | 0
Not completed — Withdrawal by Subject | 0 | 7 | 2 | 3 | 0
Not completed — Lost to Follow-up | 2 | 5 | 0 | 1 | 0
Not completed — Protocol Violation | 1 | 2 | 1 | 0 | 0
Not completed — Lack of Efficacy | 0 | 0 | 1 | 1 | 0
Not completed — Other Reason | 0 | 3 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Asthmatic Smokers Treated With Combination Therapy | Asthmatic Smoker Treated With Montelukast Only | Non-smoking Asthmatic Treated With Combination Therapy | Non-smoking Asthmatic Treated With Montelukast Only | Normal Controls | Total
Number analyzed (Participants) | 8 | 32 | 11 | 24 | 30 | 105
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 8 | 32 | 11 | 24 | 30 | 105
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 51.38 (11.41) | 36.03 (8.52) | 45.64 (17.46) | 39.00 (14.79) | 40.55 (11.35) | 40.09 (4.24)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 5 | 4 | 22 | 22 | 56
  Male | 5 | 27 | 7 | 2 | 8 | 49
Region of Enrollment [Number; unit: participants]
  Korea, Republic of | 8 | 32 | 11 | 24 | 30 | 105

OUTCOME MEASURES:

1. Secondary Outcome: Sputum Eosinophil Percentages
Description: Secondary endpoints of inflammatory markers (sputum eosinophil percentages at 24 weeks) were measured in active treatment groups
Time Frame: 24 weeks
Population: We will use ITT and PP protocols for analysis
Measure: Mean (Standard Deviation); unit: percentage of eosinophils
Arm/Group | Asthmatic Smokers Treated With Combination Therapy | Asthmatic Smoker Treated With Montelukast Only | Non-smoking Asthmatic Treated With Combination Therapy | Non-smoking Asthmatic Treated With Montelukast Only | Normal Controls
Number analyzed (Participants) | 5 | 15 | 6 | 19 | 0
percentage of eosinophils | 2.33 (3.01) | 3.60 (6.43) | 1.60 (1.34) | 3.26 (6.10) |

2. Primary Outcome: Sputum Neutrophil Percentages
Description: Week 24 sputum neutrophil percentages were measured in active treatment groups.
Time Frame: 24 weeks
Population: We will be using intention-to-treat and per protocol for analysis.
Measure: Mean (Standard Deviation); unit: percentage of neutrophils
Arm/Group | Asthmatic Smokers Treated With Combination Therapy | Asthmatic Smoker Treated With Montelukast Only | Non-smoking Asthmatic Treated With Combination Therapy | Non-smoking Asthmatic Treated With Montelukast Only | Normal Controls
Number analyzed (Participants) | 5 | 15 | 6 | 19 | 0
percentage of neutrophils | 86.00 (8.22) | 72.53 (24.14) | 89.33 (6.41) | 79.84 (17.07) |

3. Secondary Outcome: Sputum IL-8 Levels
Description: Week 24 sputum IL-8 levels in active treatment groups
Time Frame: 24 weeks
Population: We will ITT and PP protocols for analysis
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Asthmatic Smokers Treated With Combination Therapy | Asthmatic Smoker Treated With Montelukast Only | Non-smoking Asthmatic Treated With Combination Therapy | Non-smoking Asthmatic Treated With Montelukast Only | Normal Controls
Number analyzed (Participants) | 5 | 15 | 6 | 19 | 0
pg/ml | 334545 (804,831) | 26,300 (74,106) | 3602 (2342) | 317778 (738415) |

4. Secondary Outcome: Sputum GM-CSF Levels
Description: Week 24 sputum GM-CSF levels in active treatment groups were measured.
Time Frame: 24 weeks
Population: We will use ITT and PP for analysis
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Asthmatic Smokers Treated With Combination Therapy | Asthmatic Smoker Treated With Montelukast Only | Non-smoking Asthmatic Treated With Combination Therapy | Non-smoking Asthmatic Treated With Montelukast Only | Normal Controls
Number analyzed (Participants) | 5 | 15 | 6 | 19 | 0
pg/ml | 17.60 (24.67) | 15.18 (16.37) | 13.92 (10.66) | 12.16 (18.05) |

5. Secondary Outcome: Sputum IFN-gamma/IL-5 Ratios
Description: Week 24 sputum IFN-gamma/IL-5 ratios were determined in active treatment groups.
Time Frame: 24 weeks
Population: ITT and PP were used for analysis.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Asthmatic Smokers Treated With Combination Therapy | Asthmatic Smoker Treated With Montelukast Only | Non-smoking Asthmatic Treated With Combination Therapy | Non-smoking Asthmatic Treated With Montelukast Only | Normal Controls
Number analyzed (Participants) | 5 | 15 | 6 | 19 | 0
ratio | 627.4 (742.1) | 272.4 (387.1) | 183.8 (82.70) | 279.0 (563.3) |

6. Secondary Outcome: Sputum Eotaxin Levels
Description: Week 24 sputum eotaxin levels in active treatment groups were measured.
Time Frame: 24 weeks
Population: ITT and PP were used for analysis.
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Asthmatic Smokers Treated With Combination Therapy | Asthmatic Smoker Treated With Montelukast Only | Non-smoking Asthmatic Treated With Combination Therapy | Non-smoking Asthmatic Treated With Montelukast Only | Normal Controls
Number analyzed (Participants) | 5 | 15 | 6 | 19 | 0
pg/ml | 47.13 (41.93) | 87.90 (93.15) | 65.14 (25.54) | 64.61 (44.07) |

7. Secondary Outcome: Sputum RANTES Levels
Description: Week 24 sputum RANTES levels in active treatment groups were measured.
Time Frame: 24 weeks
Population: ITT and PP were used for analysis.
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Asthmatic Smokers Treated With Combination Therapy | Asthmatic Smoker Treated With Montelukast Only | Non-smoking Asthmatic Treated With Combination Therapy | Non-smoking Asthmatic Treated With Montelukast Only | Normal Controls
Number analyzed (Participants) | 5 | 15 | 6 | 19 | 0
pg/ml | 42.79 (32.47) | 44.03 (40.41) | 41.78 (19.93) | 36.41 (29.93) |

ADVERSE EVENTS:
Description: Normal Controls were not assessed for Adverse Events because they were not administered any treatment.
Arm/Group | Asthmatic Smokers Treated With Combination Therapy | Asthmatic Smoker Treated With Montelukast Only | Non-smoking Asthmatic Treated With Combination Therapy | Non-smoking Asthmatic Treated With Montelukast Only | Normal Controls
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/32 | 0/11 | 0/24 | 0/0
Other Adverse Events (participants affected / at risk) | 0/8 | 0/32 | 0/11 | 0/24 | 0/0

LIMITATIONS AND CAVEATS:
It is difficult attaining representative gender ratios (i.e., representative of the general population) when conducting a smoking study in Korea, as smoking by females is still considered culturally taboo.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No